CLINICAL TRIAL: NCT05987644
Title: DURABLE: Delayed or Upfront Brain RAdiotherapy in Treatment naïve Lung Cancer Patients With Asymptomatic or Minimally Symptomatic Brain Metastases and rEarrangements
Brief Title: Delayed or Upfront Brain RAdiotherapy in Treatment naïve Lung Cancer Patients With Asymptomatic or Minimally Symptomatic Brain Metastases and ALK rEarrangements
Acronym: DURABLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua Palmer (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joshua Palmer, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-LUN21-534
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer; NSCLC; Brain Metastases
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms | interventions — alectinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 1b: Experimental (Experimental): 600mg alectinib taken orally twice daily
  Interventions: Drug: Alectinib
- Phase 2: Arm A (Experimental): 600mg alectinib taken orally twice daily
  Interventions: Drug: Alectinib
- Phase 2: Arm B (Experimental): Subjects will receive SRS prior to taking alectinib. 24 hours after, but no more than 7 days after last radiation dose, alectinib should be taken at 600mg orally twice daily
  Interventions: Drug: Alectinib; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Alectinib — 600mg taken orally, twice daily for 25 Cycles Cycle = 4 weeks (28 days)
Radiation: Stereotactic Radiosurgery — SRS dose varies by brain met size and location
  Other Names: SRS
  Arms: Phase 2: Arm B

SUMMARY:
This study will consist of a Phase 1b and Phase 2 portion. The Phase 1b portion will enroll first followed by the Phase 2 portion. Each cycle of treatment = 28 days.

Subjects will receive alectinib twice daily. Those in the Phase 1b portion will receive alectinib alone. Those in Phase 2 Arm A will receive alectinib alone. Those in Phase 2, Arm B will receive SRS + alectinib.

A maximum of 25 cycles (2 years) of alectinib may be administered on study.

ELIGIBILITY:
General Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Fluent English skills with comprehensive/speaking skills equal to those of a native English speaker as assessed by the site investigator.
4. ECOG Performance Status of ≤ 2 within 14 days prior to registration.
5. Histological or cytological confirmation of Stage IV (per AJCC 8th edition) non-small cell lung cancer (NSCLC).
6. At least one intracranial metastasis on MRI imaging.
7. Confirmation of positive ALK rearrangement per local standard of care testing.
8. All subjects must have brain metastases and be either asymptomatic or minimally symptomatic per investigator discretion without plan for surgical intervention within 28 days of study start. Patients with neurological symptoms that are controlled with dose of corticosteroids or anti-epileptic medications are eligible. Patients with asymptomatic leptomeningeal disease may be eligible for trial providing they meet all other eligibility criteria.
9. Subjects must be planning on therapy with alectinib. Alectinib may have been started up to 6 weeks prior to registration.
10. Prior non-ALK directed therapy for metastatic disease is permitted. Patients who have received prior neoadjuvant or adjuvant chemotherapy, radiotherapy, immunotherapy (PD-1 or PD-L1 monoclonal antibodies) or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 3 months from registration since the last chemotherapy, radiotherapy, immunotherapy, or chemoradiotherapy cycle.
11. Documentation of consultation with a radiation oncologist confirming agreement to delay radiation therapy.
12. Demonstrate adequate organ function as defined in the protocol. All screening labs to be obtained within 14 days prior to registration.
13. Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. See protocol for definition of childbearing potential.
14. Females of childbearing potential and males must be willing to abstain from heterosexual intercourse or to use an effective method(s) of contraception as outlined in the protocol.
15. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
16. Patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial.
17. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

1. Active infection requiring systemic therapy.
2. Malabsorption syndrome or other condition that would interfere with enteral absorption
3. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
4. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.
5. Treatment with any investigational drug within 28 days prior to registration.
6. Acute viral, autoimmune, alcoholic, or other types of acute hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Neurological status and control of CNS disease at 12 months compared to alectinib plus SRS in patients with ≤15 CNS metastases | 12 months
  Neurological status will be measured by a composite endpoint of:
  -Inntracranial progression(icPD) by RANO-BM criteria or death during the first 12 months.
  OR
  -Symptomatic radiation necrosis during the first 12 months. Symptomatic radiation necrosis is defined as requiring initiation of or increased dose of steroids or resulting in seizures or requirement of AEDs or requirement of hospitalization or surgery.
  OR
  -Cognitive decline, defined as 1 standard deviation decline from baseline cognitive function during the first 12 months.
Phase 1b: Safety and Feasibility | 6 months
  Safety and feasibility will be assessed by frequency of Dose Limiting Toxicities.

SECONDARY OUTCOMES:
Intracranial progression-free survival at 12 months (icPFS12) | 12 months
  icPFS12 is the percentage of patients with icPD at 12 months defined by RANO-BM from randomization or death.
Intracranial disease control rate (icDCR) | 31 months
  icDCR defined as the percentage of patients with a complete response (CR), partial response (PR), or stable disease (SD), per RANO-BM.
Intracranial response rate (icRR) | 31 months
  icRR defined as the percentage of patients with a complete response (CR) and partial response (PR), per RANO-BM.
Intracranial duration of response (icDOR) | 31 months
  icDOR defined as the time when the criteria for CR or PR per RANO-BM were first met to the occurrence of an icPFS event
Extracranial PFS | 31 months
  Extracranial PFS will be defined as time from randomization to progression per RECIST v1.1
Assess Overall survival (OS) | 31 months
  OS defined as the time from randomization to death from any cause.
Safety and Tolerability | 6 months
  Safety and tolerability will be assessed by measuring the frequency and severity of adverse events based on CTCAE v5.0
Cognitive decline at 12 and 24 months | 12, 24 months
  Rate of cognitive decline, defined as 1 standard deviation decline from baseline cognitive function in at least 1 cognitive test.
Symptomatic radiation necrosis at 12 and 24 months | 12, 24 months
  Incidence of symptomatic radiation necrosis, defined as requiring initiation of or increased dose of steroids or resulting in seizures or requirement of AEDs or requirement of hospitalization or surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Palmer, MD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No